CLINICAL TRIAL: NCT00001479
Title: Intensively Sampled Dynamics of ACTH and Cortisol Affective Disorders
Brief Title: Study of the Hypothalmic-Pituitary-Adrenal (HPA) Axis and Its Role in Major Depression
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950044; 95-M-0044
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-06

CONDITIONS: Fatigue Syndrome, Chronic; Healthy; Mood Disorders
Keywords: ACTH; Adrenocorticotropic Hormone; Antidepressant Treatment; Chaos Theory; Chronic Fatigue Syndrome; Major Depression; Normal Volunteer; Primary Affective Disorder
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Mood Disorders; Depressive Disorder, Major

SUMMARY:
Major depression represents a major public health problem worldwide and in the U.S. Fifteen percent of the U.S. population has depression at some point in life (40 million individuals). The condition is more common in women, occurring at a female to male ratio of 5:2. Presently, 6-8% of all outpatients in primary care meet the diagnostic criteria for major depression. Fifteen percent of untreated patients with depression will commit suicide. Most of the people committing suicide are depressed. Researchers believe that by the year 2020 suicide will be the 10th most common cause of death in the U.S.

In addition to mortality due to suicide, depression is also associated with other severe health conditions. Areas of the brain (hippocampus) begin to deteriorate, heart disease, and decreased bone mineral density (osteoporosis) are all associated with major depression.

Researchers have believed for years that hormones controlled by the hypothalmus, pituitary gland, and adrenal gland (commonly referred to as the HPA axis or system) are in some way associated with psychiatric illnesses like depression.

According to previous studies, researchers have theorized that increased activity of the HPA axis is associated with depressed patients with typical melancholic features. Melancholia refers to the feelings of anhedonia (absence of pleasure from activites that would normally be thought of as pleasurable), insomnia (inability to sleep), guilt, and psychomotor changes. On the other hand a decrease in activity of the HPA axis may be associated with the atypical features of depression.

This study has already developed and refined studies that have improved the understanding of the HPA axis in healthy humans and depressed patients. Researchers have already identified and plan to continue identifying distinct subtypes of depressive disorders based on the activity of the HPA axis.

DETAILED DESCRIPTION:
Major depression represents a major public health problem worldwide and in the U.S. Fifteen percent of the U.S. population has depression at some point in life (40 million individuals), with a female to male ratio 5:2. Presently, 6-8% of all outpatients in primary care meet diagnostic criteria for major depression. Fifteen percent of untreated depressed patients commit suicide-most suicides have depression. In the U.S., in the year 2020 suicide will be the 10th cause of death. In addition to mortality due to suicide, major depression is associated with severe morbidity, that includes decreased hippocampal volume, cardiovascular illness, and decreased bone mineral density. Moreover, after myocardial infarction, patients with depression have a higher mortality rate than those without depression (adjusted risk ratio 4:29). Because such morbidity can be differentially affected either by increased or decreased levels of hypothalamic-pituitary-adrenal (HPA) function, it is necessary to study HPA function in our populations. Additionally, based on our previous data, we have hypothesized that depressed patients with melancholic features would have increase HPA function, while those with atypical features would have decreased HPA function. Using this protocol, over the past four years we have developed, refined, and repeatedly conducted detailed patient-oriented studies that have expanded the frontiers of existing knowledge on HPA regulation in healthy humans and depressed subjects. This protocol has already demonstrated the existence of two distinct biological subtypes of major depression, with the important finding of a decrement of HPA function in patients with atypical features. Thus, the atypical classification is not restricted to phenotype but represents a subtype with specific biological characteristics. This finding shows that there are unique strategies, targets, and potential interventional approaches to patients with either atypical or melancholic features. The elucidation of the neuroendocrinology of major depression has been a key goal of our branch, and this protocol offers the potential to unravel the biology of phenotypically distinct subtypes of major depression. Moreover, the elucidation of the medical consequences of major depression requires the precise longitudinal characterization of HPA function that is accomplished by this study.

ELIGIBILITY:
Patients with primary affective disorder (major depression), chronic fatigue syndrome, and control subjects.

Psychiatric diagnosis will be made by means of the Structured Clinical Diagnosis for DSM-III-R (SCID), performed by senior experienced clinicians.

Exclusion Criteria:

Subjects on chronic medications, which can not be washed out in one month.

Subjects with any serious medical illnesses which have been excluded.

Women who are pregnant, trying to become pregnant or sexually active and not using effective contraception.

Patients with HIV-1 infection.

Patients on chronic lithium therapy.

Subjects unable to discontinue alcohol, tobacco, or illegal drugs.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1995-01; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Babloyantz A, Destexhe A. Low-dimensional chaos in an instance of epilepsy. Proc Natl Acad Sci U S A. 1986 May;83(10):3513-7. doi: 10.1073/pnas.83.10.3513. PMID 3085091
- [Background] Demitrack MA, Dale JK, Straus SE, Laue L, Listwak SJ, Kruesi MJ, Chrousos GP, Gold PW. Evidence for impaired activation of the hypothalamic-pituitary-adrenal axis in patients with chronic fatigue syndrome. J Clin Endocrinol Metab. 1991 Dec;73(6):1224-34. doi: 10.1210/jcem-73-6-1224. PMID 1659582
- [Background] Garfinkel A, Spano ML, Ditto WL, Weiss JN. Controlling cardiac chaos. Science. 1992 Aug 28;257(5074):1230-5. doi: 10.1126/science.1519060.